CLINICAL TRIAL: NCT00527904
Title: A 12-month, Phase 3, Open-label, Multi-center Study to Evaluate the Long-term Safety of PN400 in Subjects Who Are at Risk for Developing NSAID-associated Ulcers
Brief Title: A 12-month, Phase 3, Open-label, Multi-center Study to Evaluate the Long-term Safety of PN400 (VIMOVO)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: POZEN (Industry)
Responsible Party: Senior Vice President, Clinical Research, Pozen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PN400-304
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Results first posted 2010-08-20 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Gastric Ulcer
Keywords: osteoarthritis; rheumatoid arthritis; ankylosing spondylisit; NSAIDS
MeSH Terms: conditions — Stomach Ulcer; Osteoarthritis; Arthritis, Rheumatoid | interventions — Naproxen; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PN 400 (VIMOVO) (Experimental): 500 mg delayed release naproxen/20 mg immediate release esomeprazole
  Interventions: Drug: PN400 (VIMOVO); Drug: PN 400 (VIMOVO)

INTERVENTIONS:
Drug: PN400 (VIMOVO) — Subjects are instructed to take 2 tablets a day, one in the morning and one in the afternoon/evening. The morning tablet should be taken with water, on an empty stomach 30 to 60 minutes before breakfast, or the first meal. The afternoon/evening tablet should be taken with water, on an empty stomach 30 to 60 minutes before dinner. Tablets should be swallowed whole and not broken, crushed or chewed.
  Other Names: Naprosyn; Nexium
Drug: PN 400 (VIMOVO) — 500 mg delayed-release naproxen/20 mg immediate release esomperazole dosed twice daily for 12 months
  Other Names: Naprosyn; Nexium

SUMMARY:
This study uses an open-label design and will be conducted in approximately 60 sites aiming to enroll a total number of 200 subjects to ensure that at least 100 subjects will have 12 months exposure to PN400 (VIMOVO).

DETAILED DESCRIPTION:
PN400 is proposed for the treatment of the signs and symptoms of osteoarthritis, rheumatoid arthritis and ankylosing spondylitis or other medical conditions expected to require daily NSAID therapy for at least 12 months in patients at risk for developing NSAID-associated gastric ulcers. This study is designed to provide long-term safety data for PN400 in order to gain regulatory approval to make PN400 available for clinical use in this subject population.

ELIGIBILITY:
Inclusion Criteria

A subject was eligible for inclusion in this study if all of the following criteria applied:

1. Male or non-pregnant female subjects with a history of osteoarthritis, rheumatoid arthritis, ankylosing spondylitis or other medical conditions expected to require daily NSAID therapy for at least 12 months:

   who were
   * 18-49 years of age and had a history of a documented, uncomplicated gastric or duodenal ulcer (a mucosal break of at least 3 mm in diameter with depth, without any concurrent bleeding, clot or perforation) within the past 5 years or, who were
   * 50 years of age and older (These subjects did not require a history of a documented, uncomplicated gastric or duodenal ulcer within the past 5 years).
2. Female subjects were eligible for participation in the study if they were of

   * Non-childbearing potential (i.e., physiologically incapable of becoming pregnant);
   * Childbearing potential, had negative pregnancy test at Screening, and at least 1 of the following applied or was agreed to by the subject:
   * Female sterilization or sterilization of male partner; or,
   * Hormonal contraception by oral route, implant, injectable, vaginal ring; or,
   * Any intrauterine device with published data showing that the lowest expected failure rate is less than 1% per year; or,
   * Double barrier method (2 physical barriers or 1 physical barrier plus spermicide); or
   * Any other method with published data showing that the lowest expected failure rate is less than 1% per year
3. Each subject was required to be able and willing to provide written informed consent prior to any study procedures being performed.

Exclusion Criteria

A subject was not eligible for inclusion in this study if any 1 or more of the following criteria applied:

1. History of hypersensitivity to esomeprazole or to another PPI
2. History of allergic reaction or intolerance to any NSAID (including aspirin) and/or a history of NSAID-induced symptoms of asthma, rhinitis, and/or nasal polyps
3. Participation in any study of an investigational treatment in the 4 weeks before Screening
4. Presence of uncontrolled acute or chronic medical illness, e.g., GI disorder, hypertension, diabetes, thyroid disorder, depression and/or infection that would have endangered a subject if he/she were to participate in the study
5. GI disorder or surgery leading to impaired drug absorption
6. Evidence of uncontrolled or unstable cardio- or cerebrovascular disorder which in the investigator's opinion would have endangered a subject if he/she were to participate in the study
7. Schizophrenia or bipolar disorder
8. Use of any excluded concomitant medication
9. A recent history (in the past 3 months) suggestive of alcohol or drug abuse or dependence, including overuse/abuse of narcotics for management of pain
10. Serious blood coagulation disorder, including use of systemic anticoagulants
11. Positive test result for Helicobacter pylori at Screening
12. Baseline endoscopy showing any gastric or duodenal ulcer at least 3 mm in diameter with depth
13. Screening laboratory value for any of the following tests that was > 2 times the upper limit of normal: alanine aminotransferase (ALT) and aspartate aminotransferase (AST)
14. Estimated creatinine clearance < 50 mL/min
15. Other than noted specifically, any screening laboratory value that was clinically significant in the investigator's opinion and would have endangered a subject if the subject were to participate in the study
16. History of malignancy, treated or untreated, within the past 5 years, with the exception of successfully treated basal cell or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Everardus Orlemans, PhD, Study Chair — POZEN
Locations (1):
- POZEN, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Sostek MB, Fort JG, Estborn L, Vikman K. Long-term safety of naproxen and esomeprazole magnesium fixed-dose combination: phase III study in patients at risk for NSAID-associated gastric ulcers. Curr Med Res Opin. 2011 Apr;27(4):847-54. doi: 10.1185/03007995.2011.555756. Epub 2011 Feb 14. PMID 21319944

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multi-center US study, 58 sites recruited between October 2007 and March 2009
Pre-assignment Details: Screening for eligibility and wash-out of restricted medications
Groups:
- PN400 (VIMOVO): PN 400 (20 mg esomeprazole and 500 mg naproxen) dosed twice daily
Period: Overall Study
Arm/Group | PN400 (VIMOVO)
Started | 239
Completed | 143
Not Completed | 96
Not completed — Adverse Event | 45
Not completed — Withdrawal by Subject | 21
Not completed — Lost to Follow-up | 8
Not completed — misc | 22

BASELINE CHARACTERISTICS:
Arm/Group | PN400 (VIMOVO)
Number analyzed (Participants) | 239
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 (0)
  Between 18 and 65 years | 161 (67.4)
  >=65 years | 78 (32.6)
Age Continuous [Mean (Standard Deviation); unit: years] | 60.8 (8.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168
  Male | 71
Region of Enrollment [Number; unit: participants]
  United States | 239

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Monitored for Long-term Safety of PN 400
Description: Incidence of adverse events and monitoring vital signs, clinical laboratory values, physical exams, ECG. All AEs were coded into preferred terms according to MedDRA (Medical Dictionary for Regulatory Activities) and classified by system organ class (SOC). Summaries of the incidence of all treatment-emergent AEs, treatment-related AEs, SAEs, and AEs leading to study drug discontinuation were prepared. Treatment-emergent AEs were also summarized by maximum severity, by quartile of number of doses taken and by treatment window.
Time Frame: 12 months
Population: Approximately 200 subjects were planned, 239 were enrolled and treated and 143 subjects completed the study. All 239 subjects were evaluable for safety.
Measure: Number; unit: participants
Arm/Group | PN400 (VIMOVO)
Number analyzed (Participants) | 239
participants | 239

ADVERSE EVENTS:
Time Frame: Randomization through 1 year
Arm/Group | PN400 (VIMOVO)
Serious Adverse Events (participants affected / at risk) | 13/239
Other Adverse Events (participants affected / at risk) | 175/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PN400 (VIMOVO) (N=239)
Pneumonia (Infections and infestations) | 2 (2)
Necrotizing fasciitis (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1)
Hematemesis (Gastrointestinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PN400 (VIMOVO) (N=239)
Dyspepsia (Gastrointestinal disorders) | 19 (19)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 14 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (9)
Edema peripheral (General disorders) | 11 (11)
Nausea (Gastrointestinal disorders) | 12 (12)
Abdominal pain lower (Gastrointestinal disorders) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 11 (11)
Abdominal distension (Gastrointestinal disorders) | 6 (6)
Flatulence (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 14 (14)
Bronchitis (Infections and infestations) | 9 (9)
Sinusitis (Infections and infestations) | 7 (7)
Urinary tract infection (Infections and infestations) | 6 (6)
Influenza (Infections and infestations) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5)
Headache (Nervous system disorders) | 6 (6)
Dizziness (Nervous system disorders) | 5 (5)
Contusion (Injury, poisoning and procedural complications) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Hypertension (Vascular disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees that the first publication will be a multi-center publication of the study results. Following this multi-center publication, PI can publish, present or use any non-confidential study results following Sponsor review and comment.